CLINICAL TRIAL: NCT00471731
Title: Ocular Impact of X Chromosome Karyotype and Sex Hormones in Turner Syndrome
Brief Title: Dry Eye in Women With Turner Syndrome and Women With Premature Ovarian Failure
Status: Completed | Type: Observational
Sponsor: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 070145; 07-EI-0145
Record Dates: First submitted 2007-05-09; First posted 2007-05-10 (Estimated); Last update posted 2018-02-14 (Actual); Status verified 2014-11-13

CONDITIONS: Turner Syndrome; Ovarian Failure, Premature; Sex Chromosome Aberrations; Menopause; Perimenopause
Keywords: Ocular Surface Disease; Imprinting; Eye Abnormalities; Ovarian Insufficiency; Women's Eye Health and Disease; Turner Syndrome; TS; Premature Ovarian Failure; POF; Healthy Volunteer; HV
MeSH Terms: conditions — Turner Syndrome; Primary Ovarian Insufficiency; Sex Chromosome Aberrations; Eye Abnormalities; Disease

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Premature ovarian failure (POF) is known to be associated with an increased risk of ocular surface disease (dry eye), likely due to the reduction of both estrogens and androgens seen in this condition. From preliminary data, we suspect that women with Turners syndrome (45, XO), a genetic abnormality that affects sex hormone levels, are also at increased risk of ocular surface disease. Comparing POF and TS women may allow us to distinguish different mechanisms for ocular surface disease, due to the different etiologies of hormonal (estrogen and androgen) alterations posed by POF and TS.

DETAILED DESCRIPTION:
Premature ovarian failure (POF) is known to be associated with an increased risk of ocular surface disease (dry eye), likely due to the reduction of both estrogens and androgens seen in this condition. From preliminary data, we suspect that women with Turners syndrome (45, XO), a genetic abnormality that affects sex hormone levels, are also at increased risk of ocular surface disease. Comparing POF and TS women may allow us to distinguish different mechanisms for ocular surface disease, due to the different etiologies of hormonal (estrogen and androgen) alterations posed by POF and TS.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Ability to understand and give informed consent.
  2. Meet the diagnostic criteria for TS (45, X0) or premature ovarian failure OR age matched control for study participant with TS or POF.
  3. For non Turner syndrome subjects only - Negative pregnancy test or post menopausal status for greater than or equal to 1 year.
  4. Karyotype of XO for TS subjects or XX for POF and age matched control subjects.

EXCLUSION CRITERIA:

1. Persons less than 18 years old.
2. Persons with ophthalmic diseases associated with ocular surface disease.
3. Hyperprolactinemia.
4. Cushing s syndrome.
5. Other endocrine disorders which impact sex steroid hormones.
6. AIDS
7. Pregnancy or lactation.
8. For age matched control population ONLY- complaints of dry eye.
9. For age matched control population ONLY- oral contraceptives or menopausal hormone therapy or any medications which alter sex hormone levels in the blood or chronic usage of medications that induce dry eye.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2007-05-07; Study Completion 2014-11-13

CONTACTS AND LOCATIONS:
Overall Officials: Janine A Clayton, M.D., Principal Investigator — National Eye Institute (NEI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Smith JA, Vitale S, Reed GF, Grieshaber SA, Goodman LA, Vanderhoof VH, Calis KA, Nelson LM. Dry eye signs and symptoms in women with premature ovarian failure. Arch Ophthalmol. 2004 Feb;122(2):151-6. doi: 10.1001/archopht.122.2.151. PMID 14769589
- [Background] Schaumberg DA, Buring JE, Sullivan DA, Dana MR. Hormone replacement therapy and dry eye syndrome. JAMA. 2001 Nov 7;286(17):2114-9. doi: 10.1001/jama.286.17.2114. PMID 11694152
- [Background] Coulam CB, Adamson SC, Annegers JF. Incidence of premature ovarian failure. Obstet Gynecol. 1986 Apr;67(4):604-6. PMID 3960433